CLINICAL TRIAL: NCT00266188
Title: Non-invasive Imaging and Exercise Tolerance Tests in Post-repair Tetralogy of Fallot - Intervention and Course in Patients Over 8 Years Old
Brief Title: Follow up of Post-repair Tetralogy of Fallot
Status: Completed | Type: Observational
Sponsor: Competence Network for Congenital Heart Defects (Other Government)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Other Study IDs: MP 4.1; 01G10210
Record Dates: First submitted 2005-12-15; First posted 2005-12-16 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2011-09

CONDITIONS: Tetralogy of Fallot
Keywords: Heart Defects, Congenital; Tetralogy of Fallot; Heart Septal Defects, Ventricular; Pulmonary Valve Diseases; Magnetic Resonance Imaging; Heart Catheterization; Echocardiography
MeSH Terms: conditions — Tetralogy of Fallot; Heart Defects, Congenital; Heart Septal Defects, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Tetralogy of Fallot is the most frequent complex congenital heart malformation. Over the past five decades, surgical repair has been performed with respectable results. However, relevant postoperative residues frequently remain. Pulmonary insufficiency, in particular, has been identified as a factor limiting the right ventricular function and, accordingly, the quality of life and life expectancy.

With increasing use of cardiac MRI for both measurement of ventricular function and imaging of pulmonary arteries, residual defects have been discovered that were not detectable by echocardiography. There is mounting evidence of right ventricular pressure and volume stress in Fallot patients after surgical correction. At present, it is impossible to detect right ventricular insufficiency at an early stage. Hence, it is to be assumed that right ventricular insufficiency is underdiagnosed and therapeutic action frequently is initiated beyond the point of no return of ventricular function.

The objective of this study is the systematic collection of cross-sectional and longitudinal data from extensive standardised examinations, including MRI, echocardiography, pulmonary function and ergometry tests, ECG and quality of life assessments, in a large number of patients with surgically corrected tetralogy of Fallot, and the setup of a database. The data obtained are supposed to provide information on the long-term outcome of surgical correction, to help establish criteria for necessity and time of re-intervention or re-operation, and to assess the effectiveness of re-interventions and re-operations.

DETAILED DESCRIPTION:
In the repair of tetralogy of Fallot, pulmonary insufficiency used to be tacitly accepted as a result of extensive transannular patching (TAP) and considered unobjectionable. In fact, this is well tolerated during the first postoperative years, but today there is increasing evidence that the resulting chronic volume stress to the right ventricle is harmful on the long run, in particular if there are stenoses of the pulmonary artery in addition. Such stenoses, partly due to distortions after shunt surgery, together with pulmonary insufficiency, lead to a combined volume and pressure load of the right ventricle. The chronic volume stress results in a decrease in biventricular function and exercise tolerance, associated with increasing electrical instability with frequent, mostly ventricular, dysrhythmias. This constellation brings about a significantly increased risk of cardiac death.

Pulmonary valve replacement can improve haemodynamics, exercise tolerance and dysrhythmia. However, it is still unclear, which criteria best indicate the need for re-operation or other re-intervention, such as balloon dilatations of peripheral pulmonary stenoses, and what may be the best point in time.

Cardiac MRI has been established as non-invasive method to quantify right and left ventricular function without radiation exposure. Correlating quantitative functional data to clinical conditions may permit the evaluation of factors that influence the long-term course after surgical repair of Fallot's tetralogy.

The objective of this study is to establish a broad database of cross-sectional and longitudinal (after one year) findings from extensive standardised examinations, including MRI, echocardiography, pulmonary function and ergometry tests, ECG, quality of life assessments performed and cardiac catheterisation, if indicated, on a large number of subjects with surgically corrected tetralogy of Fallot. The data obtained are supposed to determine parameters indicating beginning irreversibility of decreased cardiac function, to provide information on the long-term outcome of surgical correction, to help establish criteria for necessity and time of re-intervention or re-operation, and to assess the effectiveness of re-interventions and re-operations.

ELIGIBILITY:
Inclusion Criteria:

* Written consent of the patient and/or the patient's legal representative
* Patients with tetralogy of Fallot (including pulmonary atresia with extreme form of VSD ) after corrective operation
* The corrective intervention has to date back to at least one year before study inclusion
* Ergospirometry and MRI examination can be carried out on an outpatient basis (i. e. patients are normally older than 8 years)
* Patients are not selected according to functional status, i. e. in terms of potentially necessary reintervention measures (e. g. cardiac catheter intervention, pulmonary valve replacement)

Exclusion Criteria:

* Lack of consent
* Tetralogy of Fallot or pulmonary atresia with VSD without corrective operation (or corrective operation that dates back to less than one year before)
* Pulmonary valve agenesia, DORV (if there is a distinct discontinuity between mitral valve and aortic valve)
* Associated severe heart defects (e. g. AV canal)
* Other clinically relevant diseases, such as malignant tumour or florid diseases (in the investigating physician's assessment)
* Patient is not able to perform ergospirometry (bicycle/treadmill) or contraindication exists
* Absolute MRI contraindication, e.g. cardiac pacemaker
* Pregnant and breast-feeding patients
* Lack of cardiac catheter findings (or MRI) before initial operation -

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with tetralogy of Fallot
Sampling Method: Non-Probability Sample
Enrollment: 406 (Actual)
Dates: Start 2005-01; Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
- Assessment of the biventricular function via MRI, colour Doppler echocardiography, tissue Doppler and strain-rate imaging in correlation with objective exercise tolerance
(spiroergometry)
- Subjective quality of life
- Prevalence of cardiac dysrhythmias
- Mortality (above all in relapse interventions, such as interventional cardiac catheter or operation)
- Morbidity (i. e. severe unwanted effects [SUE], particularly in relapse interventions, such as interventional cardiac catheter or operation)

CONTACTS AND LOCATIONS:
Overall Officials: Samir Sarikouch, MD, Principal Investigator — Heart and Diabetes Center North Rhine-Westphalia; Philipp Beerbaum, MD, Study Chair — Kings College London, Division of Imaging Sciences
Locations (14):
- Germany (14):
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Deutsches Herzzentrum Muenchen, Munich, Bavaria
  - Herzzentrum Hamburg, UKE, Hamburg, Hamburg
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitätsklinikum RWTH Aachen, Aachen, North Rhine-Westphalia
  - Herz-und Diabeteszentrum Nordrhein-Westfalen, Bad Oeynhausen, North Rhine-Westphalia
  - Herzzentrum Duisburg, Duisburg, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel, North Rhine-Westphalia
  - Universitätsklinikum Muenster, Münster, North Rhine-Westphalia
  - Deutsches Kinderherzzentrum, Sankt Augustin, North Rhine-Westphalia
  - Herzzentrum Leipzig, Leipzig, Saxony
  - Deutsches Herzzentrum Berlin, Berlin, State of Berlin
  - Universitätsklinikum Charité, Berlin, State of Berlin

REFERENCES:
- [Result] Sarikouch S, Koerperich H, Dubowy KO, Boethig D, Boettler P, Mir TS, Peters B, Kuehne T, Beerbaum P; German Competence Network for Congenital Heart Defects Investigators. Impact of gender and age on cardiovascular function late after repair of tetralogy of Fallot: percentiles based on cardiac magnetic resonance. Circ Cardiovasc Imaging. 2011 Nov;4(6):703-11. doi: 10.1161/CIRCIMAGING.111.963637. Epub 2011 Sep 9. PMID 21908707
- [Result] Mueller M, Rentzsch A, Hoetzer K, Raedle-Hurst T, Boettler P, Stiller B, Lemmer J, Sarikouch S, Beerbaum P, Peters B, Vogt M, Vogel M, Abdul-Khaliq H. Assessment of interventricular and right-intraventricular dyssynchrony in patients with surgically repaired tetralogy of Fallot by two-dimensional speckle tracking. Eur J Echocardiogr. 2010 Oct;11(9):786-92. doi: 10.1093/ejechocard/jeq067. Epub 2010 May 30. PMID 20513701
- [Result] Riesenkampff E, Mengelkamp L, Mueller M, Kropf S, Abdul-Khaliq H, Sarikouch S, Beerbaum P, Hetzer R, Steendijk P, Berger F, Kuehne T. Integrated analysis of atrioventricular interactions in tetralogy of Fallot. Am J Physiol Heart Circ Physiol. 2010 Aug;299(2):H364-71. doi: 10.1152/ajpheart.00264.2010. Epub 2010 May 21. PMID 20495149
- [Result] Beerbaum P, Barth P, Kropf S, Sarikouch S, Kelter-Kloepping A, Franke D, Gutberlet M, Kuehne T. Cardiac function by MRI in congenital heart disease: impact of consensus training on interinstitutional variance. J Magn Reson Imaging. 2009 Nov;30(5):956-66. doi: 10.1002/jmri.21948. PMID 19856409
- [Result] Bodhey NK, Beerbaum P, Sarikouch S, Kropf S, Lange P, Berger F, Anderson RH, Kuehne T. Functional analysis of the components of the right ventricle in the setting of tetralogy of Fallot. Circ Cardiovasc Imaging. 2008 Sep;1(2):141-7. doi: 10.1161/CIRCIMAGING.108.783795. Epub 2008 Jul 30. PMID 19808531
- [Derived] Diller GP, Vahle J, Radke R, Vidal MLB, Fischer AJ, Bauer UMM, Sarikouch S, Berger F, Beerbaum P, Baumgartner H, Orwat S; German Competence Network for Congenital Heart Defects Investigators. Utility of deep learning networks for the generation of artificial cardiac magnetic resonance images in congenital heart disease. BMC Med Imaging. 2020 Oct 8;20(1):113. doi: 10.1186/s12880-020-00511-1. PMID 33032536
- [Derived] Orwat S, Diller GP, Kempny A, Radke R, Peters B, Kuhne T, Boethig D, Gutberlet M, Dubowy KO, Beerbaum P, Sarikouch S, Baumgartner H; German Competence Network for Congenital Heart Defects Investigators. Myocardial deformation parameters predict outcome in patients with repaired tetralogy of Fallot. Heart. 2016 Feb;102(3):209-15. doi: 10.1136/heartjnl-2015-308569. Epub 2015 Dec 29. PMID 26715570
- [Derived] Sarikouch S, Boethig D, Peters B, Kropf S, Dubowy KO, Lange P, Kuehne T, Haverich A, Beerbaum P; Investigators of the German Competence Network for Congenital Heart Defects. Poorer right ventricular systolic function and exercise capacity in women after repair of tetralogy of fallot: a sex comparison of standard deviation scores based on sex-specific reference values in healthy control subjects. Circ Cardiovasc Imaging. 2013 Nov;6(6):924-33. doi: 10.1161/CIRCIMAGING.112.000195. Epub 2013 Oct 16. PMID 24132714
- [Derived] Kutty S, Kuehne T, Gribben P, Reed E, Li L, Danford DA, Beerbaum PB, Sarikouch S. Ascending aortic and main pulmonary artery areas derived from cardiovascular magnetic resonance as reference values for normal subjects and repaired tetralogy of Fallot. Circ Cardiovasc Imaging. 2012 Sep 1;5(5):644-51. doi: 10.1161/CIRCIMAGING.112.973073. Epub 2012 Jun 22. PMID 22730421